CLINICAL TRIAL: NCT04587960
Title: Comparative Study of Outcome Between Primary Closure and Delayed Primary Closure of Skin Incision in Emergency Caesarean Section
Brief Title: Delayed Primary Closure of Skin in Emergency Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr.Jhuma Biswas (Other Government)
Responsible Party: Sponsor-Investigator, Dr.Jhuma Biswas, Associate Professor, Dept. of Obstetrics and Gynecology, Calcutta National Medical College and Hospital, Calcutta National Medical College and Hospital
Organization: Calcutta National Medical College and Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECR/771/Inst/WB/2015/RR-18
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Cesarean Wound Disruption; Cesarean Section; Infection
MeSH Terms: conditions — Infections | interventions — Cesarean Section

STUDY DESIGN:
Intervention Model Description: Patients were randomized to delayed primary closure (group A, n=40) or primary closure (group B, n=30)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary closure of Cesarean wound (Active Comparator): Immediate closure of skin incision where healing occurs by primary intention
  Interventions: Procedure: Primary closure of skin incision in Caesarean section in active comparator group
- Delayed primary closure of Cesarean wound (Experimental): Delayed closure of skin incision following regular wound dressing for 2 to 3 days.
  Interventions: Procedure: Delayed primary closure of skin incision in Caesarean section in experimental group

INTERVENTIONS:
Procedure: Delayed primary closure of skin incision in Caesarean section in experimental group — Delayed closure of skin wound of emergency Caesarean section following wound dressing for 2-3 days in experimental group
  Arms: Delayed primary closure of Cesarean wound
Procedure: Primary closure of skin incision in Caesarean section in active comparator group — Primary closure of skin wound (incisional) at the time of emergency Caesarean section in active comparator group
  Arms: Primary closure of Cesarean wound

SUMMARY:
Pregnant mothers requiring emergency cs with history of ruptured membranes would be allocated randomly into two groups in an aim to study the comparative outcome of different methods of skin closure namely primary and delayed primary closure on the incidence of wound infections requiring secondary closures and to detect the associated risk factors increasing chance of surgical site infections.

DETAILED DESCRIPTION:
OBJECTIVE

• To compare the effect of two different methods of skin wound closure namely Primary Closure and Delayed Primary Closure on the incidence of wound infection and requirement for secondary skin wound repair after emergency caesarean section in patients with ruptured membranes.

RESEARCH HYPOTHESIS Caesarean Sections (CS) in emergency situation where amniotic membrane is ruptured are clean contaminated procedures which are associated with 10-20% wound disruptions. Delayed Primary Closure for managing contaminated wounds is a concept well recognized by military surgeons, which reduces wound infections. Investigators wish to conduct this prospective study to determine the efficacy of using this technique of wound closure in Caesarean Sections in patients with history of ruptured amniotic membranes. Investigators wish to study and compare the effect of this technique versus conventional primary skin closure on wound infection and incidence of secondary wound suturing in CS with ruptured membranes.

MATERIALS AND METHODS:

1. STUDY DESIGN: Randomized controlled Trial
2. STUDY SETTING: Tertiary teaching hospital-based trial involving obstetric patients undergoing Caesarean delivery.
3. PLACE OF STUDY: Department of Obstetrics and Gynecology, Calcutta National Medical College and Hospital, Kolkata.
4. PERIOD OF STUDY: From 1st March 2020 to 15th June 2021.
5. SAMPLE SIZE: As no similar study was found in literature related to obstetric population, we have chosen an arbitrary sample size of 30 in case group and 30 in control group in this Pilot study.
6. STUDY POPULATION:

INCLUSION CRITERIA :

• Parturients admitted with rupture of membranes undergoing emergency CS

EXCLUSION CRITERIA :

* Presence of intact membranes
* Incision other than Pfannenstiel
* Presence of pre-existing infection at the site of skin incision
* Presence of obvious chorioamnionitis
* Presence of any immunosuppressive condition including HIV, intake of immunosuppressive medication, h/o chemotherapy, haematological malignancies, etc.
* Presence of other conditions interfering with wound healing like Tuberculosis, Diabetes, collagen disorders, etc.

  i) PROCEDURE:

Mothers undergoing emergency CS for various indications after rupture of membranes will be randomly allocated to two groups Study group to undergo Delayed Primary Closure of skin incision and Control group to undergo Primary closure of skin incision, after appropriate consenting.

During CS Pfannenstiel incision will be made in the skin. All patients will receive prophylactic antibiotic within thirty minutes of making abdominal incision. Depending upon the duration of membrane rupture wound will be defined either contaminated (duration of membrane rupture ≥ 12 hours) or clean contaminated (duration of membrane rupture ≤12 hours).

At the end of the procedure after closure of rectus sheath in the Study group, interrupted stitches will be taken through skin and subcutaneous tissue with 1-0 monofilament suture but knots will not be tightened and skin will be left open. Following operation, from next day onwards dressing of the wound will be done for 3 days. On 4th day, the monofilament stitches will be tightened under local anaesthesia to appose the skin. Thereafter, sutures will be removed on 7th day after operation.

In the Control group wound margins will be apposed by primary closure by interrupted stitches using 1-0 monofilament and stitches will be removed on 6th day after operation.

If there is abnormal discharge from wound, wound swabs will be taken for bacterial culture sensitivity test.

If there is wound dehiscence, timing of secondary closure will be decided based on wound health and presence of adequate granulation tissue after a period of regular wound dressing.

STASTICAL ANALYSIS PLAN Statistical methods- Linear data will be represented a mean ± standard deviation for normally distributed data and as mean (interquartile range (IQR)) for not-normally distributed data. Categorical data will represented as percentage (frequency). Comparison of means will be done with Mann Whitney U test and comparison of proportions with Chi - squared test or Fisher's exact test as appropriate. Multivariate modeling with logistic regression will be used to compare different variables between the primary closure and delayed primary closure groups.

ELIGIBILITY:
INCLUSION CRITERIA :

• Parturients admitted with rupture of membranes undergoing emergency CS

EXCLUSION CRITERIA :

* Presence of intact membranes
* Incision other than Pfannenstiel
* Presence of pre-existing infection at the site of skin incision
* Presence of obvious chorioamnionitis
* Presence of any immunosuppressive condition including HIV, intake of immunosuppressive medication, h/o chemotherapy, haematological malignancies, etc.
* Presence of other conditions interfering with wound healing like Tuberculosis, Diabetes, collagen disorders, etc.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant mothers undergoing emergency caesarean sections
Enrollment: 70 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Surgical site infections requiring secondary closure | 6 days from the day of surgery
  Incidence of surgical site infections requiring secondary closure

SECONDARY OUTCOMES:
Prolonged hospital stay | more than 7 days after surgery
  Requiring prolonged hospital stay due to wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Jhuma Biswas, MBBS, MS, Principal Investigator — Dept. of Obstetrics and Gynecology, Calcutta National Medical College and Hospital
Locations (1):
- Calcutta National Medical College and Hospital, Kolkata, West Bengal, India

IPD SHARING:
Plan to Share IPD: No
IPD would be used for this study only